CLINICAL TRIAL: NCT02773719
Title: Effect of the Intervention of Biofields Therapy on Warts of the Hands and Feet in Adults: a Prospective, Randomized, Double-blind Trial
Brief Title: Biofields Therapy on Warts
Acronym: MAGNETIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-163
Record Dates: First submitted 2016-04-22; First posted 2016-05-16 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2016-04

CONDITIONS: Wart; Energy Medecine; Magnetism
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- True biofield therapist (Experimental): Subject will have a 40 minutes therapy with a real biofield therapist to treat the wart
  Interventions: Other: True Biofield therapy
- Fake biofield therapist (Placebo Comparator): Subject will have a 40 minutes therapy with a fake biofield therapist to treat the wart
  Interventions: Other: Fake Biofield therapy

INTERVENTIONS:
Other: True Biofield therapy
  Arms: True biofield therapist
Other: Fake Biofield therapy
  Arms: Fake biofield therapist

SUMMARY:
Traditionally, healers are willing to look after, two out of three French citizens have already appealed to them at least once during their lives. Many healers in good faith are exercising their magnetism as a "gift" often inherited from elders. Now, they create interest of doctors who do not hesitate in some cases to ensure their cooperation, to implicitly recognize their mysterious talents. Some serious studies have examined these practices: Several studies have been conducted on the influence of biofield therapies in pain, depression and fatigue in cancer disease. The investigators propose a study of the effect of magnetism on the wart disease whose cure is objectively assessable.

Sixty-two subjects in total would be included, comparing 2 proportions observed: the proportion of healing in the group treated with a "real" biofield therapist (recognized and affiliated to the National Group for Alternative Medicine in France) to the proportion of healing in the group treated with a "fake" biofield therapist (someone assessed as not having capacity to magnetize). The "fake" biofield therapist, placebo, has been trained to replicate gestures during a training validated by an independent recognized biofield therapist.

ELIGIBILITY:
Patients with common warts on hands or feet for over at least 3 months are eligible for the study. Patients fulfilling one or more of the following criteria will not be included: lack of informed consent prior to randomization, younger than 18 years or under judicial protection, treated with oral corticotherapy for more than 6 months, immunosuppressed or with history of transplant surgery, undergoing chemotherapy or suspected to have carcinomatous warts, or patients with infected warts, injured warts or already treated within 90 days with chemical processing, medical device, surgery or ever treated with biofield therapy.

Subject will be excluded from the study if its warts was treated by other treatment during protocol.

* ulcerated wart
* cancerous wart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-04; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
disappearance of a common palmar or plantar wart | week 3

SECONDARY OUTCOMES:
disappearance of each other wart than the original one 3 weeks after the therapy | week 3
Percentage of reduction of each wart will be calculated using mean diameter of each wart at W0 and W3 | week3
Percentage of reduction of each wart will be calculated using mean diameter of each wart at W0 and W3 | week 3
Disappearance of warts at 6 weeks | week 6
Level of belief in biofield therapy of the subject | week 6
  week 0

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaillard C, Allain L, Legros H, Brucato S, Desgue Y, Rouillon C, Peyro-Saint-Paul L, Dompmartin A. Real versus sham proximal biofield therapy in the treatment of warts of the hands and feet in adults: study protocol for a randomized controlled trial (MAGNETIK study). Trials. 2017 Jun 7;18(1):263. doi: 10.1186/s13063-017-1994-4. PMID 28592299